CLINICAL TRIAL: NCT07397910
Title: Clinical Trial to Analyze the Effectiveness of a Natural Compound on Chronic Immune-mediated Inflammatory Status in Subjects Who Have Had SARS-CoV-2 Infection.
Brief Title: Clinical Trial on a Natural Compound to Improve Chronic Inflammation After SARS-CoV-2 Infection
Acronym: NUTRACOVID
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Bachelor of Medicine, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: UCAMCFE-00038
Record Dates: First submitted 2026-01-25; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Long COVID
Keywords: LongCOVID; Nutraceutical; Immune-inflammatory state; Exercise
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind study in relation to product consumption. Blinding cannot be performed in relation to physical exercise.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Subjects in this group will consume a placebo product (maltodextrin) with the same organoleptic characteristics as the investigational product.
  Interventions: Dietary Supplement: Control placebo; Other: No Physical Exercise
- Natural extract (Experimental): Subjects in this group will consume the investigational product (experimental product composed of a combination of six natural extracts: grapefruit extract, apigenin, orange extract, luteolin, yerba mate extract, and olive leaf extract).
  Interventions: Dietary Supplement: Experimental Product; Other: No Physical Exercise
- Physical exercise and consumption of experimental product (Experimental): During the study, subjects must consume the experimental product and also follow a training program. A multi-component program will be carried out during the 4 months of product consumption. Sessions will last 60 minutes and will be held 2-3 times per week.
  Interventions: Dietary Supplement: Experimental Product; Other: Physical exercise
- Physical exercise and consumption of placebo product (Placebo Comparator): During the study, subjects must consume the placebo product and also follow a training program. A multi-component program will be carried out during the 4 months of product consumption. Sessions will last 60 minutes and will be held 2-3 times per week.
  Interventions: Dietary Supplement: Control placebo; Other: Physical exercise

INTERVENTIONS:
Dietary Supplement: Experimental Product — Supplement consisting of orange extract, apigenin, luteolin, yerba mate extract, grapefruit extract, and olive leaf extract.
  Arms: Natural extract; Physical exercise and consumption of experimental product
Dietary Supplement: Control placebo — Product with identical characteristics to the experimental product.
  Arms: Physical exercise and consumption of placebo product; Placebo
Other: Physical exercise — During the study, subjects will have to develop a training program. A multicomponent program will be carried out during the 4 months of product consumption. The sessions will last 60 minutes and will be held 2-3 times per week.
  Arms: Physical exercise and consumption of experimental product; Physical exercise and consumption of placebo product
Other: No Physical Exercise — During the study, subjects will only consume the product assigned to them in the randomization.
  Arms: Natural extract; Placebo

SUMMARY:
A controlled, randomized clinical trial is proposed to demonstrate the effectiveness of the experimental product in controlling hepato-pulmonary inflammation and neurovascular encephalic inflammation, which may constitute the etiopathogenic basis of persistent COVID. In addition, an individualized training program will be implemented for each participant in order to improve chronic symptoms and, consequently, their quality of life.

DETAILED DESCRIPTION:
Randomized, placebo-controlled, double-blind clinical trial with four parallel arms based on the product consumed (placebo or experimental product) and the performance of physical exercise (exercise or no exercise), designed to analyze the effectiveness of the product under investigation in reducing chronic immune-mediated inflammatory status in subjects who have had SARS-CoV-2 infection and present persistent symptoms 3 months after the onset of the infectious process.

The efficacy of the experimental product, consumed over a period of 4 months, will be determined in terms of reducing chronic inflammation and improving the quality of life of people suffering from this condition.

Clinical manifestations and chronic symptoms, quality of life, response to the individualized physical exercise program, and product safety will be taken into account.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes.
* Subjects over 18 and under 70 years of age who have had a SARS-CoV-2 infection diagnosed by PDIA.
* Subjects with a history of SARS-CoV-2 infection who, three months after the onset of COVID-19, continue to experience symptoms lasting at least two months that cannot be explained by another cause. These symptoms may be newly developed after initial recovery from an acute COVID-19 episode or persist from the initial illness.
* No history of sequelae from a severe acute illness.

Exclusion Criteria:

* Subjects with an underlying disease that explains the clinical manifestations.
* Presence of chronic inflammatory diseases.
* Subjects with acute infections.
* Evidence of active thromboembolic disorder, defined as those receiving parenteral anticoagulant or thrombolytic treatment.
* Excessive alcohol consumption.
* Hypersensitivity or intolerance to any of the components of the study products.
* Use of any nutraceutical or dietary supplement.
* Severe or terminal illnesses.
* Subjects with a body mass index (BMI) over 32.
* Pregnant or lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-23 (Estimated); Primary Completion 2026-07-06 (Estimated); Study Completion 2026-08-03 (Estimated)

PRIMARY OUTCOMES:
Immunoinflammatory profile | Blood samples will be taken twice, once at baseline, at the beginning of the trial and once at the end after 120 days of product intake.
  Antibody assay for molecular biomarkers of the brain-liver-lung axis, blood-brain barrier, immunometabolic pathways, and immune-inflammatory and immuno-angiogenic cardiac remodeling.

SECONDARY OUTCOMES:
Clinical signs | It will be recorded twice, before starting the consumption of the product and before the end of consumption (120 days)
  The number of clinical manifestations, the type of manifestation, intensity according to the visual analog scale from 0 to 10, and duration of the symptomps. The clinical manifestations will be those felt by the subject.
Short Form 12 Health Survey | It will be measured twice, once at baseline and at the end of the study after 120 days of consumption.
  Measured by SF-12 questionnaire. Scale 0-100%
Sleep quality | Progress will be measured after 120 days of consumption.
  Measured by Pittsburgh test
Sleep efficiency | Progress will be measured after 120 days of consumption.
  Measured by accelerometry, with Actigraph wGT3X-BT
Fatigue | Progress will be measured after 120 days of consumption.
  Measured with Fatigue Severity Scale (FSS). Rated on a 7-point Likert scale (1=strongly disagree, 7=strongly agree), a mean score of \(\ge 4\) typically indicates a moderate to high level of fatigue.
Dyspnea | Progress will be measured after 120 days of consumption.
  It will be measured with Modified Medical Research Council (mMRC)
Depression | Progress will be measured after 120 days of consumption.
  It will be measured with Beck Depression Inventory (BDI). Scores are calculated by adding up the responses to 21 items, with a range from 0 to 63, and scores are interpreted by severity levels: 0-13 (minimal), 14-19 (mild), 20-28 (moderate), and 29-63 (severe).
Anxiety | Progress will be measured after 120 days of consumption.
  It will be measured with the State-Trait Anxiety Inventory (STAI). The STAI (State-Trait Anxiety Inventory) assesses transient (state) and stable (trait) anxiety using 40 items (20 per subscale) with a Likert-type score from 0 to 3. The total score per subscale ranges from 0 to 60, with higher scores indicating greater anxiety.
Hospital Anxiety and Depression | Progress will be measured after 120 days of consumption.
  Measured with Hospital Anxiety and Depression Scale (HADS). It is a self-administered instrument with 14 items (7 for anxiety, 7 for depression) that is scored from 0 to 3, with a maximum total of 21 points per subscale. A score of 7 or less indicates normality, 8-10 indicates a borderline case, and 11 or above indicates a probable case of anxiety or depression.
Stress level | Progress will be measured after 120 days of consumption.
  Perceived stress scale (PSS). Measures stress levels over the past month on a scale of 0 to 56. The higher the score, the greater the perceived stress. Typical interpretive ranges include low stress (0-13), moderate stress (14-26), and high stress (27-40+).
Cardiorespiratory fitness. | Progress will be measured after 120 days of consumption.
  A submaximal test will be performed.
The Rate of Force Development | Progress will be measured after 120 days of consumption.
  The Rate of Force Development (RFD) measures the speed at which the neuromuscular system generates maximum force in a short period of time (typically in the first 100-200 ms). It is a key indicator of explosive strength and power, vital in fast movements, jumps, sprints, and climbing.
Maximum Voluntary Isometric Contraction | Progress will be measured after 120 days of consumption.
  Maximum Voluntary Isometric Contraction (MVIC) is the gold standard for measuring muscle strength, involving maximum contraction without joint movement (isometric). It is used to evaluate muscle activation using electromyography, comparing the percentage of effort against the muscle's maximum possible strength.
Body composition | The test will be measured at baseline and after 16 weeks of consumption.
  It is a control variable. Measured by bioimpedance.
Liver safety variables | Hematological samples were taken before (day 0) and after consumption of the product (day 120) both in the control group and in the experimental group.
  It is a blood test that measures the presence of some enzymes, proteins and bilirubin in the blood, with the aim of determining if there is any alteration in the liver. Enzyme GPT, GOT, Gamma GT, LDH, alkaline phosphatase and bilirubin (UI/L)
Adverse events | After 16 weeks of consumption.
  It will be evaluated only at the end of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- UCAM HiTech, Sport & Health Innovation Hub, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No